CLINICAL TRIAL: NCT02486211
Title: Amantadine to Speed Awakening After Cardiac Arrest
Acronym: AWAKE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jon Rittenberger, MD (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Jon Rittenberger, MD, Associate Professor of Emergency Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15GRNT25680021
Record Dates: First submitted 2015-06-23; First posted 2015-07-01 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Coma; Heart Arrest; Anoxia
Keywords: heart arrest; resuscitation; seizures; hypothermia, induced; Amantadine
MeSH Terms: conditions — Coma; Heart Arrest; Hypoxia; Seizures; Hypothermia | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo medication administered at 0600 and 1200 via mouth, gastric tube or duo-tube.
  Interventions: Drug: Placebo
- Amantadine (Experimental): 100mg Amantadine administered at 0600 and 1200 via mouth, gastric tube or duo-tube.
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — 100mg twice per day for 7 days at 0600 and 1200
  Other Names: Symmetrel
  Arms: Amantadine
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This study evaluates if amantadine will increase the rate of awakening in patients resuscitated from cardiac arrest but comatose (not following commands) after their resuscitation. Half of the participants will receive amantadine and the other will receive placebo.

DETAILED DESCRIPTION:
Amantadine has been used to help patients awaken following traumatic brain injury, but it has not been studied in patients with anoxic brain injury.

Amantadine is a dopamine agonist and may help with stimulating the brain to awaken. The investigators will randomize subjects who remain comatose 72 hours following resuscitation from cardiac arrest to either amantadine or placebo. They will be treated with either amantadine or placebo for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Non traumatic cardiac arrest
* Age 18 and older
* Defibrillation and/or chest compressions by healthcare providers
* Return of spontaneous circulation

Exclusion Criteria:

* Written do not attempt resuscitation (DNAR) reported to providers before randomization
* Known prisoner or pregnancy
* Lack of motor response to pain and absent N20 response on somatosensory evoked potentials prior to randomization
* Initial CT demonstrating brain edema (defined as grey white ratio <1.2)
* Presence of malignant pattern on EEG at time of randomization
* Next of kin unwilling to provide supportive care for at least one week after enrollment
* Presently using other dopaminergic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon C Rittenberger, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Main Medical Center, Portland, Maine
  - Beth Israel Deacconness, Boston, Massachusetts
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amantadine | Placebo
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amantadine: 100mg Amantadine administered at 0600 and 1200 via mouth, gastric tube or duo-tube.
  Amantadine: 100mg BID for 7 days at 0600 and 1200
- Total: Total of all reporting groups
Arm/Group | Placebo | Amantadine | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9) | 54 (16) | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Rate of Awakening (Number of Patients Who Are Able to Follow Commands)
Description: Defined as the ability to follow commands (i.e. "wiggle your toes" "open your eyes" "squeeze my fingers". This corresponds to a Full Outline of Unresponsiveness motor score of 4. FOUR (full outline of unresponsiveness) measures the following: Eye Response, Motor Response, Brainstem Reflexes, and Respirations.
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 2 | 2

2. Secondary Outcome: Time to Awakening
Description: Defined as the time from enrollment to awakening
Time Frame: up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 2 | 2
days | 4 [4 to 4] | 8 [2 to 14]

3. Secondary Outcome: Seizures (Number of Patients Who Experience Seizures as Detected by EEG Monitoring With or Without Clinical Correlate)
Description: detected by EEG monitoring with or without clinical correlate
Time Frame: during study drug administration (7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 0 | 2

4. Secondary Outcome: Nausea or Vomiting
Description: nausea requiring antiemetic medications or clinical vomiting
Time Frame: during study drug administration (7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Severe or Intracranial Bleeding
Description: Bleeding that does not stop with direct pressure, requires transfusion, or occurs in the intracranial vault
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Amantadine | Placebo
All-Cause Mortality (participants affected / at risk) | 4/7 | 3/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=7) | Placebo (N=7)
Tongue swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) — Tongue swelling secondary to tongue bite.
seizure (Nervous system disorders) | 0 (0) | 2 (2) — seizure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02486211/Prot_SAP_000.pdf